CLINICAL TRIAL: NCT02544295
Title: Based-virtual Reality Diagnosis for Neuropsychiatric Diseases and Sleep/Wake Disorders
Acronym: PHENOVIRTPSY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Pierre Philip, MD / PhD, University of Bordeaux
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: UBXS 2011-02; 2011-A01418-33 (Registry Identifier: ID-RCB/EUDRACT)
Record Dates: First submitted 2015-09-03; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Aging; Addiction; Attention Deficit Disorder With Hyperactivity; Sleep Disorders; Anxiety; Depression; Attention Deficit
MeSH Terms: conditions — Behavior, Addictive; Attention Deficit Disorder with Hyperactivity; Sleep Wake Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical interview-Virtual reality task:1 (Experimental): Healthy controls will be assessed by a clinical interview by a psychiatrist, once, 1 day-duration and Virtual reality task, once, 1 day-duration
  Interventions: Behavioral: Clinical interview; Behavioral: Virtual reality task
- Clinical interview-Virtual reality task:2 (Experimental): Patients will be assessed by a clinical interview by a psychiatrist, once, 1 day-duration and Virtual reality task, once, 1 day-duration
  Interventions: Behavioral: Clinical interview; Behavioral: Virtual reality task

INTERVENTIONS:
Behavioral: Clinical interview
Behavioral: Virtual reality task

SUMMARY:
The objective of this research is to develop original virtual reality scenarios and/or new virtual reality equipments to evaluate or diagnose pathologies, such as attention deficit disorders or neuropsychiatric pathologies, addiction, anxiety or depression or pathologies interfering with sleep/wake disorders.

DETAILED DESCRIPTION:
Nature of the trial: without direct individual benefit study conducted in healthy volunteers, patients with attention disorders : ADHD (Attention Deficit Disorder / Hyperactivity) and cognitive aging, addictive disorders, anxiety disorders, depressive disorders or pathologies that interfere with sleep/wake cycle. The duration of the study is 8 years.

Type of trial: Comparison of two parallel groups of healthy volunteers and patients with attention disorders, addictive, anxious, depressive or interfering with sleep/wake cycle.

Study design:

* standardized clinical interview with a sleep specialist, psychiatrist, or psychologist and rating scales,
* a virtual reality task. The primary outcome is to evaluate the diagnosis accuracy and the acceptability of the virtual tool to the referent standard (clinical interview and scales).

The secondary outcomes are:

* The comparison of healthy subjects and patients performances
* Tolerance, acceptability to exposure to virtual scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 7 and 75 years
* Having signed written informed consent

Exclusion Criteria:

* Having participated to a clinical trial in the previous 3 months

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2012-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of the disease | 1 day
  Categorial diagnosis generated by the psychiatrist and by the Virtual reality task (0=absence of disease and 1 = presence of the disease)

SECONDARY OUTCOMES:
Sleepiness scale | 1 day
  Scores range from 0 (no sleepiness) to 24 (severe sleepiness)
BDI-II questionnaire | 1 day
  Beck Depression Inventory Scores range from 0 (no depression) to 63 (severe depression)
IDS-R questionnaire | 1 day
  Inventory of Depressive Symptomatology scores range from 0 (no depression) to 84 (severe depression)
Acceptability scale | 1 day
  Scores range from 0 to 36
ASRS | 1 day
  Adult ADHD Self-Report Scale Scores : Four or more positive answers in Part A (6 questions) are indicative of ADHD symptoms.
Physiological parameters: Polysomnography (total sleep time (min)) | 1 night
Physiological parameters: Polysomnography (sleep structure (stage %)) | 1 night
Physiological parameters: Polysomnography (Apnea/Hypopnea index and Periodic movements index (events/hr)) | 1 night

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PHILIP, PhD, Principal Investigator — University of Bordeaux
Locations (1):
- University Hospital of Bordeaux, Bordeaux, France